CLINICAL TRIAL: NCT02497001
Title: A Randomized, Double-Blind, Parallel-Group, 24-Week, Chronic-Dosing, Multi-Center Study to Assess the Efficacy and Safety of PT010, PT003, and PT009 Compared With Symbicort® Turbuhaler® as an Active Control in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Randomized, Double-Blind, Parallel-Group, 24-Week, Chronic-Dosing, Multi-Center Study to Assess the Efficacy and Safety of PT010, PT003, and PT009 Compared With Symbicort® Turbuhaler® (Kronos)
Acronym: KRONOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT010006
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BGF MDI (PT010) 320/14.4/9.6 μg ex-actuator (Experimental): BGF MDI 320/14.4/9.6 μg,Budesonide, Glycopyrronium, Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: BGF MDI 320/14.4/9.6 μg
- GFF MDI (PT003) 14.4/9.6 μg ex-actuator (Experimental): GFF MDI 14.4/9.6 μg ex-actuator Glycopyrronium, Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: GFF MDI (PT003) 14.4/9.6 μg
- BFF MDI (PT009) 320/9.6 μg ex-actuator (Experimental): BFF MDI 320/9.6 μg, Budesonide, Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: BFF MDI (PT009) 320/9.6 μg
- Symbicort (Active Comparator): Symbicort® Turbuhaler® (TBH) Inhalation Powder 200/6 μg
  Interventions: Drug: Symbicort® Turbuhaler® (TBH) Inhalation Powder

INTERVENTIONS:
Drug: BGF MDI 320/14.4/9.6 μg — Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (PT010, BGF metered dose inhaler [MDI])
  Other Names: BGF
  Arms: BGF MDI (PT010) 320/14.4/9.6 μg ex-actuator
Drug: GFF MDI (PT003) 14.4/9.6 μg — Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (PT003, GFF MDI)
  Other Names: GFF
  Arms: GFF MDI (PT003) 14.4/9.6 μg ex-actuator
Drug: BFF MDI (PT009) 320/9.6 μg — Budesonide and Formoterol Fumarate Inhalation Aerosol (PT009, BFF MDI)
  Other Names: BFF
  Arms: BFF MDI (PT009) 320/9.6 μg ex-actuator
Drug: Symbicort® Turbuhaler® (TBH) Inhalation Powder
  Arms: Symbicort

SUMMARY:
Study to Assess the Efficacy and Safety of PT010, PT003, and PT009 Compared With Symbicort® Turbuhaler® in Subjects with Moderate to Very Severe Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel-Group, 24-Week, Chronic-Dosing, Multi-Center Study to Assess the Efficacy and Safety of PT010, PT003, and PT009 Compared With Symbicort® Turbuhaler® as an Active Control in Subjects with Moderate to Very Severe Chronic Obstructive Pulmonary Disease

This study includes the following 3 sub-studies: 12-hour Pulmonary Function Test (PFT), Pharmacokinetic (PK) Profile, and Hypothalamic-pituitary-adrenal Axis.

ELIGIBILITY:
Inclusion Criteria

* Given their signed written informed consent to participate.
* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative serum pregnancy test at Visit 1, and agrees to acceptable contraceptive methods used consistently and correctly for the duration of the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS), or other local applicable guidelines.
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) ratio must be <0.70 and FEV1 must be <80% predicted normal value calculated using NHANES III reference equations (or reference norms applicable to other regions).
* Required COPD maintenance therapy:
* All Subjects must have been on two or more inhaled maintenance therapies for the management of their COPD for at least 6 weeks prior to Screening. Scheduled SABA and/or scheduled SAMA are considered inhaled maintenance therapies

Please refer to the study protocol for the complete inclusion criteria list.

Exclusion Criteria

* Significant diseases or conditions other than COPD, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening) or during the Screening Period
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening) or during the Screening Period
* Immune suppression or severe neurological disorders affecting control of the upper airway or other risk factors that in the opinion of the Investigator would put the subject at substantial risk of pneumonia.
* Subjects with a diagnosis of narrow angle glaucoma, who, in the opinion of the Investigator, have not been adequately treated.
* Subjects who have a history of hypersensitivity to β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinic anticholinergics, or any other component of the IMPs.

Please refer to the study protocol for the complete inclusion criteria list.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dorinsky, MD, Study Director — Pearl Therapeutics, Inc.
Locations (154):
- United States (57):
  - Research Site, Andalusia, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fullerton, California
  - Research Site, Gold River, California
  - Research Site, Poway, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Sacramento, California
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Dacula, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingwood, Texas
  - Research Site, Longview, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
- Canada (9):
  - Research Site, Truro, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Mirabel, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Québec
- China (27):
  - Research Site, Anqing
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Heshan
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Lianyungang
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhuhai
- Japan (61):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Date-gun
  - Research Site, Fukuoka
  - Research Site, Ginowan-shi
  - Research Site, Hakata-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiokitama-gun
  - Research Site, Higashiosaka-shi
  - Research Site, Himeji-shi
  - Research Site, Hirakata-shi
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Iwata-shi
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kahoku-gun
  - Research Site, Kakogawa-shi
  - Research Site, Kasaoka-shi
  - Research Site, Kasuga-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kiyose-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Kurashiki-shi
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsumoto-shi
  - Research Site, Matsusaka-shi
  - Research Site, Meguro-ku
  - Research Site, Mitaka-shi
  - Research Site, Mizunami-shi
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Nishishirakawa-gun
  - Research Site, Obihiro-shi
  - Research Site, Ogaki-shi
  - Research Site, Okinawa-shi
  - Research Site, Ookawa-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Ōita
  - Research Site, Ōtsu
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Seto-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Suita-shi
  - Research Site, Tachikawa-shi
  - Research Site, Takamatsu
  - Research Site, Toon-shi
  - Research Site, Toshima-ku
  - Research Site, Toyama
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Patel M, Marshall J, Martinez FJ, Mushunje A, Bowen K, Jenkins M. Frequent productive cough in COPD relates to exacerbation risk and treatment benefit from budesonide/glycopyrrolate/formoterol fumarate: a post hoc analysis of KRONOS. Respir Med. 2025 Dec;250:108499. doi: 10.1016/j.rmed.2025.108499. Epub 2025 Nov 12. PMID 41237914
- [Derived] Singh D, Bafadhel M, Arya N, Marshall J, Parikh H, Kisielewicz D, Movitz C, Bowen K, Patel M. Step up to triple therapy versus switch to dual bronchodilator therapy in patients with COPD on an inhaled corticosteroid/long-acting beta2-agonist: post-hoc analyses of KRONOS. Respir Res. 2025 May 8;26(1):175. doi: 10.1186/s12931-025-03234-5. PMID 40340809
- [Derived] Muro S, Seki M, Hurst JR, Petullo D, Marshall J, Bowen K, Darken PF, Duncan EA, Megally A, Patel M. Triple Therapy with Budesonide/Glycopyrronium/Formoterol Fumarate Dihydrate versus Dual Therapies for Patients with COPD and Phenotypic Features of Asthma: A Pooled Post Hoc Analysis of KRONOS and ETHOS. Int J Chron Obstruct Pulmon Dis. 2024 Dec 12;19:2729-2737. doi: 10.2147/COPD.S478349. eCollection 2024. PMID 39691156
- [Derived] Muro S, Kawayama T, Sugiura H, Seki M, Duncan EA, Bowen K, Marshall J, Megally A, Patel M. Benefits of budesonide/glycopyrronium/formoterol fumarate dihydrate on lung function and exacerbations of COPD: a post-hoc analysis of the KRONOS study by blood eosinophil level and exacerbation history. Respir Res. 2024 Aug 5;25(1):297. doi: 10.1186/s12931-024-02918-8. PMID 39103901
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Liu J, He X, Wu J. Economic Evaluation of Triple Therapy with Budesonide/Glycopyrrolate/Formoterol Fumarate for the Treatment of Moderate to Very Severe Chronic Obstructive Pulmonary Disease in China Using a Semi-Markov Model. Appl Health Econ Health Policy. 2022 Sep;20(5):743-755. doi: 10.1007/s40258-022-00732-1. Epub 2022 Apr 28. PMID 35478081
- [Derived] Muro S, Sugiura H, Darken P, Dorinsky P. Efficacy of budesonide/glycopyrronium/formoterol metered dose inhaler in patients with COPD: post-hoc analysis from the KRONOS study excluding patients with airway reversibility and high eosinophil counts. Respir Res. 2021 Jun 28;22(1):187. doi: 10.1186/s12931-021-01773-1. PMID 34182998
- [Derived] Huang Y, Assam PN, Feng C, Su R, Dorinsky P, Gillen M. Ethnic pharmacokinetic comparison of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler (BGF MDI) between Asian and Western healthy subjects. Pulm Pharmacol Ther. 2020 Oct;64:101976. doi: 10.1016/j.pupt.2020.101976. Epub 2020 Nov 2. PMID 33152467
- [Derived] Wang C, Yang T, Kang J, Chen R, Zhao L, He H, Assam PN, Su R, Bourne E, Ballal S, DeAngelis K, Dorinsky P. Efficacy and Safety of Budesonide/Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler in Chinese Patients with COPD: A Subgroup Analysis of KRONOS. Adv Ther. 2020 Apr;37(4):1591-1607. doi: 10.1007/s12325-020-01266-5. Epub 2020 Mar 6. PMID 32152869
- [Derived] Ichinose M, Fukushima Y, Inoue Y, Hataji O, Ferguson GT, Rabe KF, Hayashi N, Okada H, Takikawa M, Bourne E, Ballal S, DeAngelis K, Aurivillius M, Reisner C, Dorinsky P. Long-Term Safety and Efficacy of Budesonide/Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Formulated Using Co-Suspension Delivery Technology in Japanese Patients with COPD. Int J Chron Obstruct Pulmon Dis. 2019 Dec 23;14:2993-3002. doi: 10.2147/COPD.S220861. eCollection 2019. PMID 31920296
- [Derived] Dunn LJ, Kerwin EM, DeAngelis K, Darken P, Gillen M, Dorinsky P. Pharmacokinetics of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler formulated using co-suspension delivery technology after single and chronic dosing in patients with COPD. Pulm Pharmacol Ther. 2020 Feb;60:101873. doi: 10.1016/j.pupt.2019.101873. Epub 2019 Dec 10. PMID 31841699
- [Derived] Ferguson GT, Rabe KF, Martinez FJ, Fabbri LM, Wang C, Ichinose M, Bourne E, Ballal S, Darken P, DeAngelis K, Aurivillius M, Dorinsky P, Reisner C. Triple therapy with budesonide/glycopyrrolate/formoterol fumarate with co-suspension delivery technology versus dual therapies in chronic obstructive pulmonary disease (KRONOS): a double-blind, parallel-group, multicentre, phase 3 randomised controlled trial. Lancet Respir Med. 2018 Oct;6(10):747-758. doi: 10.1016/S2213-2600(18)30327-8. Epub 2018 Sep 16. PMID 30232048
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4148&filename=PT010006-02_FINAL_Redacted_17MAY2018.pdf
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010006&attachmentIdentifier=e464d4a5-e38a-47b1-8e03-b8acd1cbd842&fileName=PT010006_SAP_v2.0_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 208 sites in four countries, from August 2015 until January 2018. The entire study period could take up to a maximum of 30 weeks.
Pre-assignment Details: Subjects were randomized in a 2:2:1:1 scheme.
Groups:
- BGF MDI 320/14.4/9.6 ug: Budesonide Glycopyrronium Formoterol Fumarate Metered Dose Inhalation 320/14.4/9.6 ug
- GFF MDI 14.4/9.6 ug: Glycopyrronium Formoterol Fumarate Metered Dose Inhalation 14.4/9.6 ug
- BFF MDI 320/9.6 ug: Budesonide Formoterol Fumarate Metered Dose Inhalation 320/9.6 ug
- Symbicort TBH 400/12 ug: Symbicort Turbuhaler 400/12 ug
Period: Overall Study
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug
Started | 640 | 627 | 316 | 319
Completed | 566 | 524 | 266 | 278
Not Completed | 74 | 103 | 50 | 41
Not completed — Lost to Follow-up | 10 | 2 | 0 | 2
Not completed — Adverse Event | 28 | 30 | 11 | 11
Not completed — Withdrawal by Subject | 14 | 37 | 19 | 15
Not completed — Physician Decision | 5 | 11 | 5 | 1
Not completed — subjects that were not treated | 1 | 2 | 2 | 1
Not completed — Major Protocol Deviation | 3 | 4 | 4 | 4
Not completed — Lack of Efficacy | 10 | 16 | 6 | 6
Not completed — Protocol Violation | 3 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: mITT - Modified Intent to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug | Total
Number analyzed (Participants) | 639 | 625 | 314 | 318 | 1896
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: mITT
  Years | 64.9 (7.8) | 65.1 (7.7) | 65.2 (7.2) | 65.9 (7.7) | 65.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 195 | 90 | 82 | 546
  Male | 460 | 430 | 224 | 236 | 1350
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT
  Participants
    Hispanic or Latino | 16 | 14 | 7 | 4 | 41
    Not Hispanic or Latino | 623 | 611 | 305 | 312 | 1851
    Unknown or Not Reported | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Asian | 284 | 285 | 142 | 141 | 852
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
    Black or African American | 23 | 38 | 15 | 14 | 90
    White | 329 | 301 | 157 | 163 | 950
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-4
Description: FEV1 AUC0-4 (L) for The Efficacy Estimand (Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve from 0 to 4 hours (AUC0-4) AUC was normalized for length of follow up (e.g. typically 4 hours)).
Time Frame: at Week 24
Population: mITT population total numbers may vary based on predefined subject exclusions prior to study unblinding
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Symbicort®: Symbicort® Turbuhaler® (TBH) Inhalation Powder
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 436 | 403 | 201 | 211
Liters | 0.292 [0.271 to 0.314] | 0.288 [0.266 to 0.310] | 0.177 [0.146 to 0.207] | 0.189 [0.160 to 0.219]

2. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Description: Morning Pre-Dose Trough FEV1 (L) for The Efficacy Estimand
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 565 | 522 | 266 | 276
Liters | 0.124 [0.108 to 0.140] | 0.111 [0.094 to 0.127] | 0.050 [0.027 to 0.072] | 0.062 [0.039 to 0.084]

3. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Description: Morning Pre-Dose Trough FEV1 (L) for The Efficacy Estimand
Time Frame: over 24 Weeks
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 622 | 601 | 300 | 301
Liters | 0.147 [0.134 to 0.159] | 0.125 [0.112 to 0.137] | 0.073 [0.055 to 0.091] | 0.088 [0.070 to 0.105]

4. Secondary Outcome: Peak Change From Baseline in FEV1 Within 4 Hours Post-dosing
Description: Peak Change from Baseline in FEV1 (L) Within 4 Hours Post-Dose for The Efficacy Estimand
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 436 | 403 | 201 | 211
Liters | 0.370 [0.348 to 0.393] | 0.361 [0.338 to 0.384] | 0.253 [0.221 to 0.284] | 0.264 [0.233 to 0.295]

5. Secondary Outcome: Rate of Moderate or Severe COPD Exacerbations
Description: Rate of Moderate or Severe COPD Exacerbations for the Efficacy Estimand
Time Frame: over 24 weeks
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: Exacerbations
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 108 | 157 | 65 | 61
Exacerbations | 0.46 (0.05) | 0.95 (0.09) | 0.56 (0.08) | 0.55 (0.08)

6. Secondary Outcome: Percentage of Subjects Achieving a Minimal Clinically Important Difference (MCID) of 4 Units or More in SGRQ Total Score (SGRQ Responders)
Description: Change from BGF
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 625 | 314 | 318
Percentage | 6.06 [0.30 to 11.82] | 6.43 [-0.62 to 13.47] | 8.23 [1.23 to 15.22]

7. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin HFA Use
Description: Change from Baseline in Mean Daily Number of Puffs of Rescue Ventolin HFA for The Efficacy Estimand
Time Frame: over 24 Weeks
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 141 | 155 | 269 | 233
Puffs | -1.3 [-1.6 to -1.1] | -1.1 [-1.3 to -0.8] | -1.1 [-1.5 to -0.8] | -1.6 [-1.9 to -1.2]

8. Secondary Outcome: Time to Onset of Action on Day 1, 5 Minutes Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 429 | 417 | 220 | 210
Liters | 0.181 [0.169 to 0.192] | 0.194 [0.182 to 0.205] | 0.167 [0.152 to 0.182] | 0.163 [0.148 to 0.178]

9. Secondary Outcome: Time to Onset of Action on Day 1, 15 Minutes Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 484 | 470 | 238 | 238
Liters | 0.217 [0.205 to 0.230] | 0.230 [0.218 to 0.243] | 0.197 [0.180 to 0.213] | 0.190 [0.174 to 0.207]

10. Secondary Outcome: Time to Onset of Action on Day 1, 30 Minutes Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 490 | 474 | 242 | 238
Liters | 0.236 [0.223 to 0.249] | 0.255 [0.242 to 0.268] | 0.213 [0.195 to 0.230] | 0.208 [0.190 to 0.225]

11. Secondary Outcome: Time to Onset of Action on Day 1, 1 Hour Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 497 | 481 | 244 | 245
Liters | 0.268 [0.254 to 0.282] | 0.282 [0.268 to 0.296] | 0.228 [0.208 to 0.247] | 0.232 [0.213 to 0.251]

12. Secondary Outcome: Time to Onset of Action on Day 1, 2 Hours Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 494 | 480 | 243 | 246
Liters | 0.281 [0.266 to 0.295] | 0.292 [0.277 to 0.307] | 0.241 [0.220 to 0.261] | 0.244 [0.224 to 0.265]

13. Secondary Outcome: Time to Onset of Action on Day 1, 4 Hours Post Dose
Description: FEV1 (L) by Post-Dose Timepoint on Day 1 for The Efficacy Estimand
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | BGF MDI 320/14.4/9.6 μg | GFF MDI (PT003) 14.4/9.6 μg | BFF MDI (PT009) 320/9.6 μg | Symbicort®
Number analyzed (Participants) | 491 | 477 | 243 | 244
Liters | 0.276 [0.260 to 0.292] | 0.278 [0.262 to 0.294] | 0.234 [0.213 to 0.256] | 0.247 [0.225 to 0.268]

ADVERSE EVENTS:
Time Frame: Serious Adverse events were collected from the time subject signed Informed Consent to the time of the final follow-up telephone call. Adverse Events were collected from the time subject was randomized.
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least 1 dose of the study drug.
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug
All-Cause Mortality (participants affected / at risk) | 6/639 | 3/625 | 2/314 | 1/318
Serious Adverse Events (participants affected / at risk) | 55/639 | 68/625 | 21/314 | 29/318
Other Adverse Events (participants affected / at risk) | 126/639 | 84/625 | 59/314 | 55/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=639) | GFF MDI 14.4/9.6 ug (N=625) | BFF MDI 320/9.6 ug (N=314) | Symbicort TBH 400/12 ug (N=318)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 32 (41) | 8 (8) | 13 (16)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 6 (6) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue ferver (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitits (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metasteses of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metasteses to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischeamia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Siezure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident6 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delerium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=639) | GFF MDI 14.4/9.6 ug (N=625) | BFF MDI 320/9.6 ug (N=314) | Symbicort TBH 400/12 ug (N=318)
Nasopharyngitits (Infections and infestations) | 49 (61) | 41 (48) | 26 (30) | 30 (32)
Upper Respiratory Infection (Infections and infestations) | 65 (77) | 37 (41) | 18 (18) | 22 (23)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 21 (21) | 8 (9) | 17 (18) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02497001/SAP_000.pdf
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02497001/Prot_001.pdf